CLINICAL TRIAL: NCT06756594
Title: Efficacy of Dexmedetomidine-Propofol Versus Ketamine-Propofol for Sedation During Gastrointestinal Endoscopy
Brief Title: Efficacy of Dexmedetomidine-Propofol Versus Ketamine-Propofol for Sedation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Hany Hamed, Resident, Department of Anesthesia, Intensive Care and Pain management, Faculty of Medicine, Sohag University, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Soh-Med-24-11-02MS
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-11

CONDITIONS: Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dexmedetomidine-Propofol for sedation during gastrointestinal endoscopy (Active Comparator): efficacy of sedation with Dexmedetomidine-Propofol combination in the upper or lower gastrointestinal system endoscopy.
  Interventions: Drug: Dexmedetomidine-Propofol
- Ketamine-Propofol for sedation during gastrointestinal endoscopy (Active Comparator): efficacy of sedation with Ketamine-Propofol combination in the upper or lower gastrointestinal system endoscopy.
  Interventions: Drug: Ketamine-Propofol

INTERVENTIONS:
Drug: Dexmedetomidine-Propofol — efficacy of sedation with Dexmedetomidine-Propofol combination in the upper or lower gastrointestinal system endoscopy.
  Arms: Dexmedetomidine-Propofol for sedation during gastrointestinal endoscopy
Drug: Ketamine-Propofol — efficacy of sedation with Ketamine-Propofol combination in the upper or lower gastrointestinal system endoscopy.
  Arms: Ketamine-Propofol for sedation during gastrointestinal endoscopy

SUMMARY:
This study aims to compare efficacy of sedation between Dexmedetomidine-Propofol and Ketamine-Propofol combinations in the upper or lower gastrointestinal system endoscopy. We compare between 2 combinations as regard hemodynamic stability, post operative side effects as occurrence of delirium, nausea, vomiting, headache, hallucination or agitation.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I to II.
* Age between 18 and 60 years.
* Both sexes.

Exclusion Criteria:

* Having severe heart, lung, liver disease, kidney failure, or bleeding disorder.
* Patients having fever, hypothermia or infection, electrolyte disorders, such as hypokalemia and hypocalcaemia, acid-base disorder, allergy to drugs to be used.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2025-06-11 (Estimated); Study Completion 2025-06-11 (Estimated)

PRIMARY OUTCOMES:
intraoperative and postoperative monitoring of sedation during upper or lower gastrointestinal system endoscopy. | every 5 minutes intraoperative and every 15 minutes for 2 hours postoperative.
  Sedation level

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] Tekeli AE, Oguz AK, Tuncdemir YE, Almali N. Comparison of dexmedetomidine-propofol and ketamine-propofol administration during sedation-guided upper gastrointestinal system endoscopy. Medicine (Baltimore). 2020 Dec 4;99(49):e23317. doi: 10.1097/MD.0000000000023317. PMID 33285707
- [Background] Zhang F, Sun HR, Zheng ZB, Liao R, Liu J. Dexmedetomidine versus midazolam for sedation during endoscopy: A meta-analysis. Exp Ther Med. 2016 Jun;11(6):2519-2524. doi: 10.3892/etm.2016.3186. Epub 2016 Mar 24. PMID 27284342
- [Background] Chang ET, Certal V, Song SA, Zaghi S, Carrasco-Llatas M, Torre C, Capasso R, Camacho M. Dexmedetomidine versus propofol during drug-induced sleep endoscopy and sedation: a systematic review. Sleep Breath. 2017 Sep;21(3):727-735. doi: 10.1007/s11325-017-1465-x. Epub 2017 Jan 27. PMID 28130737